CLINICAL TRIAL: NCT04256915
Title: A Randomised Controlled Trial of the Effects of Cognitive Behavioural Therapy and Bright Light Therapy for Insomnia in Adolescents With Evening Chronotype
Brief Title: Effects of Cognitive Behavioural Therapy and Bright Light Therapy for Insomnia in Adolescents With Evening Chronotype
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Chinese University of Hong Kong (Other); University of Oxford (Other); Flinders University (Other)
Responsible Party: Principal Investigator, Dr. Shirley Xin Li, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EA1802063
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Insomnia; Delayed Sleep Phase
Keywords: Insomnia; Eveningness; Adolescents; Youth; Light therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy; Ultraviolet Therapy

STUDY DESIGN:
Intervention Model Description: For both treatment groups, the intervention will consist of 6 weekly sessions of cognitive behavioural therapy for insomnia (CBT-I) (90-min, 3-6 adolescents in each group). Participants in both groups will be also instructed to undergo morning light therapy (by wearing Re-timers) at home for 30 minutes daily. Re-timers can be worn like a pair of glasses, with 2 light-emitting diodes (LEDs) per eye. The following two conditions will be delivered by Re-timers: participants in the CBT-I group will receive a placebo light intervention where they will be exposed to dim red light (50lux), whereas participants in the CBT-I plus light therapy group will receive the active light treatment, with 2 LEDs emitting constant diffused blue-green light (500 nm, 506 lux).
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CBT-I + Bright Light (Experimental): n = 50
  Interventions: Behavioral: Cognitive Behavioural Therapy for Insomnia (CBT-I) + Bright Light Therapy
- CBT-I + Placebo Light (Active Comparator): n = 50
  Interventions: Behavioral: Cognitive Behavioural Therapy for Insomnia (CBT-I) + Placebo Light Therapy
- Wait-list Control (No Intervention): n = 50

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy for Insomnia (CBT-I) + Bright Light Therapy — CBT-I consists of 6 weekly sessions of CBT-I (90-min, 3-6 adolescents in each group) with elements that address the behavioural, cognitive and physiological factors perpetuating insomnia, including: psycho-education about sleep and sleep hygiene, stimulus control, sleep restriction, relaxation training, structured worry time, cognitive restructuring (targeting sleep-related dysfunctional cognitions), and relapse prevention.
  Participants will additionally undergo daily morning light therapy by wearing Re-timers (a validated portable light emitting device) at home for 30 minutes. Participants will receive constant blue-green light (500 nm, 506 lux).
  Arms: CBT-I + Bright Light
Behavioral: Cognitive Behavioural Therapy for Insomnia (CBT-I) + Placebo Light Therapy — CBT-I consists of 6 weekly sessions of CBT-I (90-min, 3-6 adolescents in each group) with elements that address the behavioural, cognitive and physiological factors perpetuating insomnia, including: psycho-education about sleep and sleep hygiene, stimulus control, sleep restriction, relaxation training, structured worry time, cognitive restructuring (targeting sleep-related dysfunctional cognitions), and relapse prevention.
  Participants will additionally undergo daily morning light therapy by wearing Re-timers (a validated portable light emitting device) at home for 30 minutes.Participants will receive red-filtered dim light (<50 lux).
  Arms: CBT-I + Placebo Light

SUMMARY:
Insomnia is prevalent in adolescents. Together with an increase of evening preference (i.e. evening chronotype) in adolescent, sleep disturbance in adolescents are associated with a constellation of adverse outcomes. Insomnia and evening chronotype in adolescents are also found to predict the development of mental health problems and negative health-related outcomes in young adulthood.

While cognitive behavioural therapy for insomnia (CBT-I) and bright light therapy were evidenced to be effective in managing sleep problems in adults, there is limited evidence to support their efficacy in children and adolescents. To address the limitations in the existing literature, this study aims to conduct a randomised controlled trial to examine the effects of CBT-I and light therapy on insomnia and mood symptoms, and other clinical and daytime symptoms, as well as overall functioning in adolescents with insomnia (particularly sleep onset insomnia) and evening chronotype.

DETAILED DESCRIPTION:
A randomised, assessor-blind, parallel group controlled trial will be conducted in youth with insomnia and eveningness. Eligible participants will be randomised to one of the following groups: CBT-I, CBT-I plus bright light therapy, or waiting-list control. Randomisation will be carried out using an automated online system. Assessments will be conducted at pre-treatment (week 0), during the treatment (week 2 & 4) and post-treatment (week 6/at the conclusion of the last group session). The two active treatment groups will be additionally followed up at post-treatment one-month and post-treatment six months in order to examine the maintenance effects following the intervention with CBT-I and CBT-I plus bright light therapy respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese aged 12-24 years old;
2. Predominant complaint of difficulty in initiating sleep at least three times a week and for at least 3 months;
3. Show clinically significant impairment / distress;
4. Having a score of >= 9 on the Insomnia Severity Index (ISI) ;
5. Classified as evening chronotype based on the score of reduced Horne-Östberg Morning-Eveningness Questionnaire (rMEQ; i.e. <12) and having a sleep onset time of 11:15pm or later for 12 year olds, 11:30pm or later for 13-14 year olds, and 12:00am or later for 15 years or above at least 3 nights per week for the past 3 month as confirmed by a 7-day sleep diary;
6. Written informed consent of participation into the study is given by the participant and his/her parent or guardian (for those aged under 18);
7. Being able to comply with the study protocol.

Exclusion Criteria:

1. Current diagnosis of substance abuse or dependence; current or history of manic or hypomanic episode, schizophrenia spectrum disorders, neurodevelopmental disorders, organic mental disorders, or intellectual disabilities;
2. Having a prominent medical condition known to interfere with sleep continuity and quality (e.g. eczema);
3. Having a clinically diagnosed sleep disorder that may potentially contribute to a disruption in sleep continuity and quality (e.g. narcolepsy) as ascertained by the Structured Diagnostic Interview for Sleep Patterns and Disorder (DISP);
4. Concurrent, regular use of medications known to affect sleep continuity and quality;
5. Initiation of and change of medication that may interfere with circadian rhythm within past 3 months (e.g. lithium);
6. In the opinion of the research clinician, having a clinically significant suicidality (presence of suicidal ideation with a plan or an attempt);
7. Currently receiving any other structured psychotherapy;
8. With hearing or speech deficit;
9. Presence of an eye disease (e.g. retinal blindness);
10. Night shift worker;
11. Trans-meridian flight in the past 3 months and during the study.

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Insomnia Symptoms | Baseline, Post-Treatment (at the conclusion of the last session) for all participants, and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Insomnia symptoms measured by Insomnia Severity Index (ISI). ISI is a 5-item self-rated scale. Possible scores range from 0 to 20, with higher scores indicating higher insomnia severity.

SECONDARY OUTCOMES:
Change in Sleep Quality | Baseline, Post-Treatment (at the conclusion of the last session) for all participants, and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Pittsburgh Sleep Quality Index (PSQI) is a self-rated scale consisting of 19 questions. All items are combined to form seven component scores on different aspects of sleep quality, each of which ranges from 0 to 3 points with higher scores representing more sleep disturbance. The seven component scores are added to one global score, which ranges from 0 to 21, with higher scores indicating more difficulties with sleep.
Change of Sleep Diary Measure - Time in Bed (TIB) | Baseline, Post-Treatment (at the conclusion of the last session) for all participants, and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: time in bed (TIB) in hours
Change of Sleep Diary Measure - Total Sleep Time (TST) | Baseline, Post-Treatment (at the conclusion of the last session) for all participants, and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: total sleep time (TST) in hours
Change of Sleep Diary Measure - Sleep Onset Latency (SOL) | Baseline, Post-Treatment (at the conclusion of the last session) for all participants, and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: sleep onset latency (SOL) in mins
Change of Sleep Diary Measure - Wake After Sleep Onset (WASO) | Baseline, Post-Treatment (at the conclusion of the last session) for all participants, and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: wake after sleep onset (WASO) in mins
Change of Sleep Diary Measure - Sleep Efficiency (SE) | Baseline, Post-Treatment (at the conclusion of the last session) for all participants, and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: sleep efficiency (SE), which is calculated by total sleep time divided by total time in bed, %
Change in Objective Sleep Measures - Time in Bed (TIB) | Baseline, Post-Treatment (at the conclusion of the last session) for all participants, and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Actigraphic assessment for consecutive seven days. Sleep parameter estimated by wrist actigraphy: time in bed (TIB) in hours
Change in Objective Sleep Measures - Total Sleep Time (TST) | Baseline, Post-Treatment (at the conclusion of the last session) for all participants, and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Actigraphic assessment for consecutive seven days. Sleep parameter estimated by wrist actigraphy: total sleep time (TST) in hours
Change in Objective Sleep Measures - Sleep Onset Latency (SOL) | Baseline, Post-Treatment (at the conclusion of the last session) for all participants, and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Actigraphic assessment for consecutive seven days. Sleep parameter estimated by wrist actigraphy: sleep onset latency (SOL) in mins
Change in Objective Sleep Measures - Wake After Sleep Onset (WASO) | Baseline, Post-Treatment (at the conclusion of the last session) for all participants, and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Actigraphic assessment for consecutive seven days. Sleep parameter estimated by wrist actigraphy: wake after sleep onset (WASO) in mins
Change in Objective Sleep Measures - Sleep Efficiency (SE) | Baseline, Post-Treatment (at the conclusion of the last session) for all participants, and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Actigraphic assessment for consecutive seven days. Sleep parameter estimated by wrist actigraphy: sleep efficiency (SE), which is calculated by total sleep time divided by total time in bed, %
Change in Self-Report Chronotype Measures | Baseline, Post-Treatment (at the conclusion of the last session) for all participants, and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  The Munich Chronotype Questionnaire (MCTQ) is a self-report measures of sleeping patterns during weekdays and weekends separately. The Mid-Sleep Time (MSF/MSFsc) are used to as an indicator of chronotype, where individuals with earlier mid-sleep time reflect a morning chronotype and later mid-sleep time reflect an evening chronotype.
Change in Actigraphic Circadian Measures using Nonparametric circadian rhythm analysis - interdaily stability (IS) | Baseline, Post-Treatment (at the conclusion of the last session) for all participants, and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Actigraphic assessment for consecutive seven days. Circadian parameters computed by the nonparametric circadian rhythm analysis method - interdaily stability (IS), which is calculated as the ratio between the variance of the average 24-hour pattern around the mean and the overall variance.
Change in Actigraphic Circadian Measures using Nonparametric circadian rhythm analysis - intradaily variability (IV) | Baseline, Post-Treatment (at the conclusion of the last session) for all participants, and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Actigraphic assessment for consecutive seven days. Circadian parameters computed by the nonparametric circadian rhythm analysis method - intradaily variability (IV), which is calculated as the ratio of the mean squares of the difference between consecutive hours and the mean squares around the grand mean.
Change in Actigraphic Circadian Measures using Nonparametric circadian rhythm analysis - M10 | Baseline, Post-Treatment (at the conclusion of the last session) for all participants, and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Actigraphic assessment for consecutive seven days. Circadian parameters computed by the nonparametric circadian rhythm analysis method - start times and average activity of M10 (i.e. 10 h with maximal activity).
Change in Actigraphic Circadian Measures using Nonparametric circadian rhythm analysis - L5 | Baseline, Post-Treatment (at the conclusion of the last session) for all participants, and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Actigraphic assessment for consecutive seven days. Circadian parameters computed by the nonparametric circadian rhythm analysis method - start times and average activity of L5 (i.e. five hours with least activity).
Change in Actigraphic Circadian Measures using Nonparametric circadian rhythm analysis - relative amplitude (RA) | Baseline, Post-Treatment (at the conclusion of the last session) for all participants, and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Actigraphic assessment for consecutive seven days. Circadian parameters computed by the nonparametric circadian rhythm analysis method - relative amplitude (RA), which is calculated using L5 and M10 to give a nonparametric description of amplitude.
Change in Actigraphic Circadian Measures using Cosinor Analysis - acrophase | Baseline, Post-Treatment (at the conclusion of the last session) for all participants, and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Actigraphic assessment for consecutive seven days. Circadian parameters computed by the cosinor analysis method - acrophase (the peak of the sine wave).
Change in Actigraphic Circadian Measures using Cosinor Analysis - amplitude | Baseline, Post-Treatment (at the conclusion of the last session) for all participants, and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Actigraphic assessment for consecutive seven days. Circadian parameters computed by the cosinor analysis method - amplitude (the difference between the wave peak and trough).
Change in Actigraphic Circadian Measures using Cosinor Analysis - mesor | Baseline, Post-Treatment (at the conclusion of the last session) for all participants, and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Actigraphic assessment for consecutive seven days. Circadian parameters computed by the cosinor analysis method - mesor.
Change in Objective Circadian Measures: Dim-light melatonin onset (DLMO) | Baseline, Post-Treatment (at the conclusion of the last session) for all participants
  Dim-light melatonin onset (express as time value hh:mm) is determined by 10-hours salivary melatonin collected at 30-minutes interval. Melatonin is assayed by gas chromatography-mass spectrometry.
Change of Depressive Symptoms (Assessor-rated) | Baseline, Post-Treatment (at the conclusion of the last session) for all participants, and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Children's Depression Rating Scale (CDRS-R) is a 17-item rating scale based on a semistructured interview with children. Possible scores range from 17 to 113, with higher scores indicating severer depressive symptoms.
Change of Self-report Mood Symptoms | Baseline, Post-Treatment (at the conclusion of the last session) for all participants, and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Hospital Anxiety and Depression Scale (HADS) is a self-assessed scale for detecting states of depression and anxiety. The depression subscale range in scores from 0 to 21, with higher scores indicating severer states of depression. Similarly, the anxiety subscale range in scores from 0-21 with higher scores indicating severer states of anxiety. No additional computation will be made with the two subscores.
Change of Suicidal Ideation | Baseline, Post-Treatment (at the conclusion of the last session) for all participants, and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Depressive Symptom Inventory Suicidality Subscale (DSI-SS) is a 4-item self-rated scale measuring suicidal ideation. Possible total scores range from 0 to 12, with higher scores indicating higher suicidal ideation.
Change of Daytime Sleepiness | Baseline, Post-Treatment (at the conclusion of the last session) for all participants, and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Paediatric Daytime Sleepiness Scale (PDSS) is an 8-item self-rated scale measuring daytime sleepiness, ranging in total scores from 0 to 32 with higher scores indicating more sleepiness.
Change of Daytime Fatigue | Baseline, Post-Treatment (at the conclusion of the last session) for all participants, and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Multidimensional Fatigue Inventory (MFI) is a 20-item self-rated scale on fatigue symptoms. There are three subscales, measuring the physical (possibly scored from 7 to 35), mental (possibly scored from 6 to 30), and spiritual (possibly scored from 7 to 35), dimensions of fatigue. A grand total score can be calculated by summing up the three sub scores. In all cases, a higher score represents higher fatigue symptoms.
Change of Quality of Life (KIDSCREEN-27) | Baseline, Post-Treatment (at the conclusion of the last session) for all participants, and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  KIDSCREEN-27 is a 27-item self-rated scale measuring health related quality of life measure for children and adolescents. There are five subscales on: physical well-being (possibly scored from 5 to 25), psychological well-being (possibly scored 7 to 35), autonomy & parents (possibly scored 7 to 35), peers & social support (possibly scored 4 to 20), and school environment (possibly scored 4 to 20). A grand total score can be calculated by summing up the five sub scores. In all cases, a higher score represents higher perceived well-being.
Change of Overall Severity of Clinical Symptoms | Baseline, Post-Treatment (at the conclusion of the last session) for all participants, and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Clinical Global Impression (CGI) Scale is a clinician-rated scale, comprised of two one-item subscales: Severity of Illness (CGI-S) subscale evaluating the severity of psychopathology, and Clinical Global Improvement Scale (CGI-I) evaluating change from the initiation of treatment. In both cases, the score is given on a seven-point scale, with higher values indicating higher severity of illness and larger improvement respectively.
Change of Objective Cognitive Performance (visual attention & task switching) | Baseline, Post-Treatment (at the conclusion of the last session) for all participants, and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Trail Making Test for assessing visual attention and task switching. In Trail Making Test, longer reaction time indicates lower level of attention.
Change of Objective Cognitive Performance (inhibitory ability) | Baseline, Post-Treatment (at the conclusion of the last session) for all participants, and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Go/No-go Task for assessing inhibitory ability. In Go/No-go Task, a higher error rate indicates lower inhibition control.
Change of Objective Cognitive Performance (working memory by digit span) | Baseline, Post-Treatment (at the conclusion of the last session) for all participants, and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Digit Span Task for assessing working memory capacity. In Digit Span Task, a higher number of recalled digits indicates better working memory.
Change of Objective Cognitive Performance (working memory by N-Back) | Baseline, Post-Treatment (at the conclusion of the last session) for all participants, and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  N-back Task for assessing working memory capacity and manipulation. In N-back Task, a d prime score will be calculated based on the signal detection theory, where a higher score indicates better working memory performance.
Change of Objective Cognitive Performance (episodic memory) | Baseline, Post-Treatment (at the conclusion of the last session) for all participants, and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Chinese Auditory Verbal Learning Task for assessing episodic memory, where a higher number of recalled words indicates better episodic memory performance.
Change of Objective Cognitive Performance (problem solving) | Baseline, Post-Treatment (at the conclusion of the last session) for all participants, and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Wisconsin Card Sorting Test for assessing problem solving. In Wisconsin Card Sorting Test, lower executive functioning is indicated by a higher percentage of persistent errors and a higher number of trials taken to complete the first category.
Change of sleep related attention bias | Baseline, Post-Treatment (at the conclusion of the last session) for all participants, and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Sleep-related Dot-Probe Task for assessing sleep-related attention bias. In the Sleep-related Dot-probe Task, a higher attention bias score indicates higher vigilance towards sleep-related stimuli.
Change of risk-taking & decision making | Baseline, Post-Treatment (at the conclusion of the last session) for all participants, and additional two follow-ups at Post-Treatment 1-month and Post-Treatment 6-month for participants in the treatment groups
  Balloon Analogue Risk Task for assessing risk-taking and decisionmaking. In Balloon Analogue Risk Task, a score will be calculated by averaging the number of pumps on unexploded blue balloons, where a higher score indicates more risk-taking and impulsive propensities.

CONTACTS AND LOCATIONS:
Locations (1):
- Sleep Research Clinic and Laboratory, Department of Psychology, The University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Li SX, Cheung FTW, Chan NY, Chan JWY, Zhang J, Li AM, Espie CA, Gradisar M, Wing YK. Effects of cognitive behavioural therapy and bright light therapy for insomnia in youths with eveningness: study protocol for a randomised controlled trial. Trials. 2024 Apr 9;25(1):246. doi: 10.1186/s13063-024-08090-0. PMID 38594725